CLINICAL TRIAL: NCT04281823
Title: Houston Methodist DeBakey Cardiovascular Magnetic Resonance Study
Brief Title: DeBakey Cardiovascular Magnetic Resonance Study
Acronym: DEBAKEY-CMR
Status: Recruiting | Type: Observational
Sponsor: Dipan Shah (Other)
Responsible Party: Sponsor-Investigator, Dipan Shah, Director of Cardiovascular Imaging, The Methodist Hospital Research Institute
Organization: The Methodist Hospital Research Institute (Other)
Other Study IDs: Pro00008766
Record Dates: First submitted 2020-01-24; First posted 2020-02-24 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Cardiovascular Diseases
Keywords: Cardiovascular Disease; Cardiac Magnetic Resonance; Myocardial Fibrosis; Valvular Heart Disease; Ischemic Heart Disease; Cardiomyopathy
MeSH Terms: conditions — Cardiovascular Diseases; Heart Valve Diseases; Myocardial Ischemia; Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiovascular Magnetic Resonance: All patients who present to the Houston Methodist CMR Laboratory
  Interventions: Diagnostic Test: Cardiovascular Magnetic Resonance

INTERVENTIONS:
Diagnostic Test: Cardiovascular Magnetic Resonance — Patients will undergo various CMR techniques designed to assess cardiovascular structure and function, tissue characteristics, and flow.

SUMMARY:
While advancements in cardiac magnetic resonance (CMR) have improved image quality, it is unclear how these improvements are connected to the clinical evaluation of individuals with cardiovascular disease. The aim of this large prospective registry revolves around 4 key principles: 1) utilize CMR to gain additional pathophysiologic insights into cardiovascular disease, 2) understand how CMR compares to alternative cardiovascular diagnostic modalities, 3) determine how CMR affects clinical management decisions, and 4) establish a link between CMR findings and long term prognosis in patients with known or suspected cardiovascular disease. The ultimate aim is to utilize CMR to improve patient outcomes.

CMR techniques to be studies include function, fibrosis, and flow. Focus areas include valvular heart disease, ischemic heart disease, cardiomyopathies, and vascular disease.

DETAILED DESCRIPTION:
Patient Population, Recruitment, and Consent:

Patients presenting to the Houston Methodist DeBakey CMR Laboratory will be enrolled from April 2008 to April 2038. It is expected that up to 100,000 patients may be enrolled during this period.

Subjects will be identified based on their referral to the Houston Methodist DeBakey CMR Laboratory for MRI studies during the proposed study period.

After enrollment, a registered nurse or physician will perform a thorough structured patient interview and/or review of electronic health records to document baseline medical history including cardiac risk factors, symptoms, medication usage, and prior procedure history. A small blood sample will be drawn and stored for future biomarker and/or genetic testing analysis. Annual follow up for clinical status will be performed via review of electronic health records; structured telephone interviews with the patients, relatives, and/or their health care providers; and/or the social security death index database.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting to the Houston Methodist CMR Laboratory with known or suspected cardiovascular disease.

Exclusion Criteria:

* Unable to provide informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: All patients present to the Houston Methodist CMR Laboratory providing informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2008-04-01 (Actual); Primary Completion 2058-04-01 (Estimated); Study Completion 2058-04-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | Through study completion, an average of once a year, up to 20 years
  All-cause mortality, Cardiovascular mortality (acute Myocardial Infarction, sudden death, heart failure, cerebrovascular, procedural), and Non-cardiovascular mortality
Heart Failure | Through study completion, an average of once a year, up to 20 years
  Congestive heart failure
Heart and/or Lung Transplantation | Through study completion, an average of once a year, up to 20 years
Left Ventricular and/or Right Ventricular Assist Device Implantation | Through study completion, an average of once a year, up to 20 years

SECONDARY OUTCOMES:
Cardiac Interventions | Through study completion, an average of once a year, up to 20 years
  Implantable cardioverter-defibrillator (ICD), pacemakers, cardiac resynchronization therapy, coronary revascularization, valvular intervention, shunt closure
Arrhythmic | Through study completion, an average of once a year
  Sustained ventricular tachycardia, ventricular fibrillation, nonfatal cardiac arrest, appropriate ICD therapy
Acute myocardial infarction | Through study completion, an average of once a year, up to 20 years
Acute Cerebrovascular Accident | Through study completion, an average of once a year, up to 20 years

CONTACTS AND LOCATIONS:
Overall Officials: Dipan Shah, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Participant data will not be made available to other researchers.

REFERENCES:
- [Derived] Tayal B, Faza NN, Nguyen DT, Malahfji M, Little S, Saeed M, Goel SS, Guha A, El-Tallawi KC, Graviss EA, Shah DJ. Association of secondary mitral regurgitation and right ventricular dysfunction among patients with non-ischaemic cardiomyopathy. Eur Heart J Cardiovasc Imaging. 2024 Nov 27;25(12):1627-1635. doi: 10.1093/ehjci/jeae134. PMID 38781428
- [Derived] Tayal B, Debs D, Nabi F, Malahfji M, Little SH, Reardon M, Zoghbi W, Kleiman N, Shah DJ. Impact of Myocardial Scar on Prognostic Implication of Secondary Mitral Regurgitation in Heart Failure. JACC Cardiovasc Imaging. 2021 Apr;14(4):812-822. doi: 10.1016/j.jcmg.2020.11.004. Epub 2020 Dec 16. PMID 33341417
- [Derived] Kitkungvan D, Yang EY, El Tallawi KC, Nagueh SF, Nabi F, Khan MA, Nguyen DT, Graviss EA, Lawrie GM, Zoghbi WA, Bonow RO, Quinones MA, Shah DJ. Extracellular Volume in Primary Mitral Regurgitation. JACC Cardiovasc Imaging. 2021 Jun;14(6):1146-1160. doi: 10.1016/j.jcmg.2020.10.010. Epub 2020 Dec 16. PMID 33341409